CLINICAL TRIAL: NCT06878560
Title: EXPAND: A Prospective Study to Evaluate the Safety and Efficacy of the 10 GE Xenokidney in Patients With End-stage Renal Disease (ESRD)
Brief Title: Study to Evaluate the Safety and Efficacy of the 10 GE Xenokidney in Patients With ESRD
Acronym: EXPAND
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPK-KF-101
Record Dates: First submitted 2025-03-03; First posted 2025-03-17 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: ESRD (End-Stage Renal Disease); Kidney Transplantation; Xenotransplantation
Keywords: 10 GE Xenokidney; End-stage renal disease; ESRD; Xenotransplantation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: This single group study will enroll participants simultaneously from either of two patient populations: (1) participants that are ineligible for conventional allogeneic kidney transplantation due to medical reason or (2) participants on an Organ Procurement and Transplantation Network kidney transplant waitlist that are more likely to die or go untransplanted within 5 years than receive a kidney transplant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 10 GE Xenokidney (Experimental): Participants will receive 10 GE Xenokidney
  Interventions: Biological: 10 GE Xenokidney

INTERVENTIONS:
Biological: 10 GE Xenokidney — Porcine-derived kidney containing intentional genomic alterations for xenotransplantation
  Other Names: Xenokidney; UKidney

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the 10 GE Xenokidney in patients with ESRD who are either not eligible for conventional allogeneic kidney transplantation (Group 1) or are on an Organ Procurement and Transplantation Network (OPTN) kidney transplant waitlist, but are more likely to die or go untransplanted within 5 years than receive a kidney transplant (Group 2).

The study consists of xenotransplantation followed by a 24-week Post-transplant Follow up Period (Part A) to evaluate the efficacy and safety objectives followed by a Long-term Follow-up Period (Part B) to evaluate participant survival, 10 GE Xenokidney survival, and screening for zoonotic infections. Part B will continue for the lifetime of the participant.

DETAILED DESCRIPTION:
This is a Phase 1/2/3, multicenter, open-label, safety and efficacy study of the 10 GE Xenokidney in patients with ESRD. The study will be comprised of the following:

* A Screening Period up to 52 weeks.
* Part A consists of the 10 GE Xenokidney transplantation followed by a 24-week Post-transplant Follow-up Period, including the evaluation of all study endpoints and safety assessments.
* Part B is a Long-term Follow-up Period that extends for the lifetime of participants who received the 10 GE Xenokidney, including but not limited to documentation of participant survival, 10 GE Xenokidney survival, and screening for zoonotic infections.

There will be 2 groups of participants enrolled in the study. Group 1 will be participants deemed ineligible for conventional allogeneic kidney transplantation due to medical reason(s). Group 2 will be participants on an OPTN kidney transplant waitlist but are more likely to die or go untransplanted within 5 years than receive a kidney transplant.

ELIGIBILITY:
Inclusion Criteria for all Participants (Groups 1 and 2):

1. Provide voluntarily informed consent to participate in the study and for lifetime follow up.
2. Have a diagnosis of ESRD at the time of informed consent.
3. Hemodialysis dependent for a minimum of 6 months and has a functioning arterial venous fistula/graft or permanent catheter at the time of informed consent.
4. 50 to 70 years of age at the time of informed consent, or 40 to <50 years of a age with a calculated panel reactive antibody (cPRA) of ≥99.9%.
5. Live withing 3 hours travel time of the xenotransplant center.
6. Female participants must be postmenopausal or permanently sterilized (eg, hysterectomy, bilateral oophorectomy, or bilateral salpingectomy). Male participants must agree to the use of a highly effective method of birth control, if the possibility of conception exists.
7. Negative xeno-crossmatch at Screening and pre-transplant.
8. Estimated Post Transplant Survival Calculator score >20% (https://optn.transplant.hrsa.gov/data/allocation-calculators/epts-calculator/).
9. Body mass index ≤35 kg/m2.
10. Have completed or have initiated and plan to complete (meningococcal A, C, W, Y and meningococcal B vaccine series only) Centers for Disease Control and Prevention recommended courses of age and risk factor appropriate vaccinations.
11. Seropositive (immunoglobulin G) for cytomegalovirus and Epstein-Barr virus.

Additional Inclusion Criteria for Group 1:

1. Ineligible for conventional allogeneic kidney transplantation due to medical reason(s) for any of the following:

1. Ineligible for a living donor transplant.
2. Ineligible for an OPTN kidney transplant waitlist (reason for ineligibility will be collected).
3. Delisted from OPTN kidney transplant waitlist (reason for delisting will be collected).

Additional Inclusion Criteria for Group 2:

1. On an OPTN kidney transplant waitlist (active or inactive status).
2. No approved living kidney donors.
3. More likely to die or go untransplanted within 5 years than receive a kidney transplant as measured by the Kidney Transplant Decision Aid at the time of informed consent (select United States for "Choose your state" field and National average for "Choose your transplant program" field; https://www.srtr.org/tools/kidney-transplant-decision-aid/).

Exclusion Criteria (pertain to all participants in Groups 1 and 2):

1. Need for multiple organ transplants.
2. Severe medical co-morbidities including, but not limited to:

   1. Chronic liver disease.
   2. Advanced cardiovascular disease.
   3. Severe peripheral vascular disease that limits technical ability to transplant the 10 GE Xenokidney.
   4. Severe neurologic diseases or conditions that would preclude meaningful recovery or informed consent.
   5. Oral steroid-dependent airway disorder or chronic pulmonary disease or requires chronic, intermittent or continuous supplemental oxygen.
   6. Pulmonary hypertension.
   7. Uncontrolled diabetes or sequelae of diabetes mellitus including severe non-proliferative diabetic retinopathy.
   8. Severe neurogenic bladder that requires intermittent catheterization.
3. ESRD due to hereditary or structural kidney disease.
4. Active or recently treated malignancy at the time of informed consent.
5. Non-renal cause of hematological disorders associated with anemia (eg, thalassemia and sickle disease).
6. Cannot discontinue chronic anticoagulation therapy (low-dose daily aspirin is permissible).
7. History of major psychiatric disorders with a psychiatric hospitalization and/or suicidal ideation within 5 years of informed consent.
8. Being treated for active tuberculosis (TB), have received prophylaxis for positive FDA-approved interferon-gamma release assay, or test positive for TB by FDA-approved interferon-gamma release assay test during Screening.
9. Nucleic acid test (NAT) positive for hepatitis B virus and/or hepatitis C virus, hepatitis B surface antibody (anti HBs) titer <10 mIU/mL unless the participant is determined to be a nonresponder to hepatitis B vaccination (a nonresponder is defined as having an anti-HBs titer <10 mIU/mL after having completed both the standard vaccine series and a fourth booster dose and/or second standard vaccine series), and/or positive for human immunodeficiency virus (HIV; HIV-1 and HIV-2 antibody and/or NAT).
10. Not able to independently perform activities of daily life.
11. Have a history of medical noncompliance that may preclude adherence to the demands and requirements of xenotransplantation (eg, history of substance use disorder (SUD) within 1 year of informed consent, lack of social support, untreated psychological conditions).

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2075-10 (Estimated)

PRIMARY OUTCOMES:
Survival Rate of Patients with ESRD Receiving the 10 GE Xenokidney at 24 Weeks Post Transplant | Day 0 (day of xenotransplantation) to 24 weeks post transplant
  Participant survival rate at 24 weeks post transplant.
Survival Rate of the 10 GE Xenokidney at 24 Weeks Post Transplant | Day 0 (day of xenotransplantation) to 24 weeks post transplant
  10 GE Xenokidney survival rate at 24 weeks post transplant. 10 GE Xenokidney failure is defined as 10 GE Xenokidney nephrectomy.
Survival Time of Participants Receiving the 10 GE Xenokidney | Day 0 (day of xenotransplantation) until death for any cause, assessed at least every 24 weeks after transplantation while the participant is alive, up to 50 years
  Participant survival post transplant. Participant survival is defined as time from xenotransplantation to death for any cause
Survival Time of the 10 GE Xenokidney (Overall Survival) | Day 0 (day of xenotransplantation) until start of chronic dialysis, nephrectomy, or death, whichever occurs first, assessed at least every 24 weeks after transplantation while the participant is alive and the xenokidney is functional, up to 50 years
  Overall survival of the 10 GE Xenokidney post transplant. Overall survival time of the 10 GE Xenokidney is defined as time from xenotransplantation to 10 GE Xenokidney nephrectomy or death, whichever occurs first.
Survival Time of the 10 GE Xenokidney (Death-censored Survival) | Day 0 (day of xenotransplantation) until start of chronic dialysis, nephrectomy, or death, whichever occurs first, assessed at least every 24 weeks after transplantation while the participant is alive and the xenokidney is functional, up to 50 years
  Death-censored survival 10 GE Xenokidney. Death-censored survival time of the 10 GE Xenokidney is defined as time from xenotransplantation to 10 GE Xenokidney nephrectomy censored for death.
10 GE Xenokidney Function Post Transplant (Endogenous GFR) | At 24 weeks post transplant
  Endogenous measured GFR (24-hour urine creatinine clearance) at 24 weeks post transplant.
10 GE Xenokidney Function Post Transplant (Exogenous GFR) | At 24 weeks post transplant
  Exogenous measured GFR (nuclear medicine GFR) at 24 weeks post transplant.
Quality of Life in Participants Receiving the 10 GE Xenokidney by EuroQol 5-Dimension 5-Level (EQ-5D-5L) | Baseline to 24 weeks post transplant
  Change in the EQ-5D-5L from baseline to 24 weeks post transplant. The EQ-5D-5L questionnaire assesses health-related quality of life across 5 categories (Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression).
  Each category has 5 levels, ranging from 1 (no problems) to 5 (extreme problems or inability to perform the activity). Higher scores indicate a worse health outcome (more mobility issues, greater pain, more anxiety, etc).
Quality of Life in Participants Receiving the 10 GE Xenokidney by Standardized Outcomes in Nephrology Life Participant (SONG-LP) | Baseline to 24 weeks post transplant
  Change in SONG-LP from baseline to 24 weeks post transplant. The SONG-LP assesses participation in different life activities over the past month. The minimum score (worst outcome) is 4 (if all responses are "1" - Never) and the maximum score (best outcome) is 20 (if all responses are "5" - Always). Higher scores indicate a better health outcome (greater ability to participate in activities).
Quality of Life in Participants Receiving the 10 GE Xenokidney by Kidney Transplant Questionnaire (KTQ) | Baseline to 24 weeks post transplant
  Change in KTQ from baseline to 24 weeks post transplant. Each question in the KTQ is scored on a 1 to 7 scale with: 1 = worst outcome (eg, "A very great deal of trouble or distress" / "All of the time") and 7 = best outcome (eg, "No trouble or distress" / "None of the time"). Higher scores indicate a better outcome, meaning less distress, fewer symptoms, and better well-being.
Quality of Life in Participants Receiving the 10 GE Xenokidney by Patient Global Impression of Change (PGI-C) | At 24 weeks post transplant
  PGI-C at 24 weeks post transplant. The PGI-C assesses a patient's perception of improvement or worsening over time. The minimum score (best outcome) is 1 ("Very Much Improved") and the maximum score (worst outcome) is 7 ("Very Much Worse"). Higher scores indicate a worse health outcome (greater worsening).
Incidence of Treatment-Emergent Adverse Events (Safety of the 10 GE Xenokidney) | Baseline until last visit, assessed at least every 24 weeks after transplantation while the participant is alive and the xenokidney is functional, up to 50 years, or for 1 year after nephrectomy if required
  Incidence of adverse events and serious adverse events; all-cause mortality.
Incidence of Proteinuria | Day 0 (day of xenotransplantation) until last visit, assessed at least every 24 weeks after transplantation while the participant is alive and the xenokidney is functional, up to 50 years, or for 1 year after nephrectomy if required
  Incidence of proteinuria from Day 0.
Incidence of Zoonotic Infection | Day 0 (day of xenotransplantation) until last visit, assessed at least every 24 weeks after transplantation while the participant is alive and the xenokidney is functional, up to 50 years, or for 1 year after nephrectomy if required
  Incidence of zoonotic infection from Day 0.
Incidence of Opportunistic Infection | Day 0 (day of xenotransplantation) until last visit, assessed at least every 24 weeks after transplantation while the participant is alive and the xenokidney is functional, up to 50 years, or for 1 year after nephrectomy if required
  Incidence of opportunistic infection from Day 0.

CONTACTS AND LOCATIONS:
Locations (1):
- New York University Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No